CLINICAL TRIAL: NCT01101568
Title: A Study to Investigate the Interaction of GSK1292263 With Rosuvastatin and Simvastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113506
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GSK1292263, rosuvastatin, simvastatin, pharmacokinetics, drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Simvastatin; Rosuvastatin Calcium; (1-(3-isopropyl-1,2,4-oxadiazol-5-yl)piperidin-4-yl)methyl methanesulfonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Sequence (Experimental): Simvastatin will be administered on Day 1 and Day 10. Rosuvastatin will be administered on Day 3 and Day 12. GSK1292263 will be administered on Days 6 to 14.
  Interventions: Drug: Simvastatin; Drug: Rosuvastatin; Drug: GSK1292263

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40mg (single dose) on Days 1 and 10.
Drug: Rosuvastatin — Rosuvastatin 10mg (single dose) on Days 3 and 12.
Drug: GSK1292263 — GSK1292263 300mg BID Days 6 to 14.

SUMMARY:
This study is a Phase I, open-label, single-sequence drug interaction study to evaluate the effect of repeated doses of GSK1292263 on the pharmacokinetics of rosuvastatin and simvastatin in healthy adult subjects. Each subject will receive single doses of simvastatin and rosuvastatin on two occasions, once alone and once following administration of repeated (BID) doses of GSK1292263.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or bilateral oophorectomy or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. If the clinical situation is unclear, FSH and estradiol levels may be used to confirm post-menopausal status at Screening. Simultaneous follicle stimulating hormone (FSH) > 40 mIU/ml and estradiol < 40pg/ml (<140pmol/L) is confirmatory in the absence of a clear post-menopausal history.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 5 terminal half-lives (i.e. 4 days) post-last dose.
* Body weight greater than or equal to 50 kg and BMI within the range 19 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Subjects with cholelithiasis or obstructive or inflammatory gallbladder disease within 3 months prior to Screening are excluded.
* Gastrointestinal disease that could affect fat or bile acid absorption, or the pharmacokinetics or pharmacodynamics of the study drugs, including inflammatory bowel disease, chronic diarrhea, Crohn's or malabsorption syndromes within the past year
* Gastrointestinal surgery that may affect the pharmacokinetics or pharmacodynamics of the study drugs
* Subjects may be enrolled in the study if they have had a cholecystectomy three or more months before the time of screening and are stable and asymptomatic.
* Significant ECG abnormalities, defined in the protocol. Subjects with Left Bundle Branch Block are excluded from the study. Subjects with partial Right Bundle Branch Block may be considered for inclusion following consultation with the GSK Medical Monitor. Subjects with WPW syndrome are excluded from the study.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma, (e.g., for any FTIH where risk of bronchoconstriction is unknown, or compound specific where risk of bronchoconstriction).
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* CPK above the upper limit of normal at screening.
* Lactose intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04-14 (Actual); Primary Completion 2010-06-24 (Actual); Study Completion 2010-06-24 (Actual)

PRIMARY OUTCOMES:
AUC(0-inf) and Cmax of rosuvastatin alone and in the presence of GSK1292263 | Day 3 and Day 12
AUC(0-inf) and Cmax of simvastatin/simvastatin acid alone and in the presence of GSK1292263 | Day 1 and Day 10

SECONDARY OUTCOMES:
Safety and tolerability: adverse events, cardiovascular findings (blood pressure, heart rate, ECGs) and clinical laboratory values. | Throughout the study (Day 1 to Day 25)
PK parameters: time to maximum plasma concentration, apparent plasma terminal elimination half-life and area under the plasma concentration-time curve for rosuvastatin [AUC(0-72 hours)] and simvastatin/simvastatin acid [AUC(0-24h)] | 15 days
PK parameter values: AUC(0-24h), Cmax, tmax and t1/2 for GSK1292263 and assessment of steady-state | From Day 6 to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113506 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113506?search=study&study_ids=113506#rs
- Available data/document: Clinical Study Report: 113506 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113506 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113506 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113506 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113506 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113506 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113506 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register